CLINICAL TRIAL: NCT06020664
Title: A Randomized, Placebo Controlled, Evaluator-Blinded Study to Assess the Efficacy and Safety of NOX1416 in the Treatment of Chronic, Non-Healing, Diabetic Foot Ulcers
Brief Title: NOX1416 in Treatment of Chronic Non-Healing Diabetic Foot Ulcers (NTCDU)
Acronym: NTCDU
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: The NO-002 study had to be paused because of enrollment disruptions due to the current situation in Israel, and concerns over the placebo batch stability results.
Sponsor: NOxy Health Products, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NO-002
Record Dates: First submitted 2023-07-10; First posted 2023-08-31 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: A total of 30 subjects will be randomized 1:1 to receive either NOX1416 + SOC or Placebo + SOC (15 per group).
Who Masked: Outcomes Assessor
Masking Description: Evaluator-Blinded Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NOX1416+SOC (Experimental): NOX1416 is a foam based gaseous nitric oxide (NO) product that will be topically applied directly onto the wound bed and left on the wound bed for a 5-minute period. Subjects randomized to the NOX1416 treatment group will receive once a day application, for a total of 12 weeks with a double treatment, 10 minutes apart, on the first day. Standard of care will include evaluation to document, off-loading adequate arterial flow, wound cleaning, removal of necrotic, infected and/or nonviable tissue by debridement, maintenance of moist wound environment, and management of infection.
  Interventions: Drug: NOX-1416+SOC
- Placebo+SOC (Placebo Comparator): Placebo is topically applied directly onto the wound bed and left on the wound bed for a 5-minute period. Subjects randomized to the control group will receive once a day application, for a total of 12 weeks with a double treatment, 10 minutes apart, on the first day. Standard of care will include evaluation to document, off-loading adequate arterial flow, wound cleaning, removal of necrotic, infected and/or nonviable tissue by debridement, maintenance of moist wound environment, and management of infection.
  Interventions: Other: Placebo+SOC

INTERVENTIONS:
Drug: NOX-1416+SOC — NOX1416+SOC as provided in Arm/group description
  Other Names: Advanox
  Arms: NOX1416+SOC
Other: Placebo+SOC — Placebo+SOC as provided in Arm/group description
  Arms: Placebo+SOC

SUMMARY:
The goal of this multi-center,randomized, placebo controlled, evaluator-blinded study is to assess the efficacy and safety of NOX1416 in the treatment of chronic, non-healing, diabetic foot ulcers (DFUs). Subjects will be randomized to receive treatment with NOX1416 or placebo as an adjunct to SOC.

The primary objective of the study is to evaluate the clinical benefit of daily NOX1416, as an adjunct to standard of care (SOC), in the treatment of chronic, non-healing DFUs. The secondary objective is to demonstrate efficacy, safety and tolerability of NOX1416 as adjunct to SOC. Each site will assign a physician (or designee) to serve as the "blinded-evaluator" to be responsible for assessing the study endpoints such as wound measurements and complete wound closure. The blinded-evaluator will not be involved in the clinical care of the subject.

DETAILED DESCRIPTION:
A total of 30 subjects will be randomized 1:1 to receive either NOX1416 + SOC or Placebo + SOC. NOX1416 is a foam based gaseous nitric oxide (NO) product where NO is delivered through a microbubble foam. One pump each of Solution A (0.3g, containing Citric acid) and Solution B (0.3g, containing Sodium nitrite) will be dispensed, mixed for five seconds and applied immediately per each square centimeter of wound area using any sterile applicator. NOX1416 is topically applied directly onto the wound bed and left on the wound bed for a 5-minute period.

Subjects randomized to the NOX1416 treatment group will receive once a day application, for a total of 12 weeks with a double treatment, 10 minutes apart, on the first day. Similar to the NOX1416 treatment schedule, placebo will be topically applied directly onto the wound bed and left on the wound bed for a 5-minute period. Subjects randomized to the control group will receive once a day application, for a total of 12 weeks with a double treatment, 10 minutes apart, on the first day.

Standard of care will include evaluation to document, off-loading adequate arterial flow, wound cleaning, removal of necrotic, infected and/or nonviable tissue by debridement, maintenance of moist wound environment, and management of infection.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for enrollment in the study only if they meet ALL the following criteria at time of Screening:

1. Male or female subjects aged 18 to 80 years (inclusive) with Type 1 or Type 2 diabetes undergoing therapy for glycemic control.
2. Subject has a glycosylated hemoglobin, HbA1c ≤ 12%. Note: Prior documented HbA1c within the last 3 months of the Screening Visit is acceptable.
3. Presence of at least one diabetic foot ulcer that meets all of the following criteria:

   1. A full-thickness ulcer of University of Texas Wound Classification (UTWCS) Grade I or II
   2. Ulcer is located on or below the malleoli
   3. Ulcer size (area) is ≥ 1 cm2 and ≤ 10 cm2 (post-debridement at time of randomization)
   4. Unresponsive to standard ulcer care and present for ≥1 month and ≤1 year (at time of screening)
   5. There is a minimum 1 cm margin between the qualifying Target Ulcer and any other ulcers on the specified foot, post-debridement)
   6. No exposed bone and no tunneling, undermining, or sinus tracts
   7. Ulcer must be non-healing as defined as <35% reduction in size in response to standard of care during the two-week run-in Screening Period (between the first Screening Visit and Baseline) Note: Criterion 3(g) will be evaluated at the time of randomization. If the subject has more than one qualifying diabetic foot ulcer, the ulcer designated as the Target Ulcer will be at the discretion of the Investigator.
4. Subject has adequate vascular perfusion of the affected limb, confirmed by Ankle-Brachial Index (ABI) ≥ 0.6 and ≤ 1.2. ABI results within the last 3 months of Screening are acceptable. The assessment may also be performed between SV1 and SV2.

   Note: If the ABI measurement is >1.20, confirmatory tests (Great toe pressure and/or TcPO2 at the foot) will be performed. A subject will be considered eligible for inclusion in this study if Great toe pressure ≥ 40mmHg or TcPO2 ≥ 40 mmHg at the foot. Prior documented flow study within the last 3 months of the Screening Visit is acceptable.
5. Clinically normal resting ECG at Screening Visit or, if abnormal, considered not clinically significant by the Principal Investigator.
6. Subject, if female of child-bearing potential, has a negative serum pregnancy test at screening, must not be breastfeeding, and willing to use acceptable methods of contraception (birth control pills, barriers, or abstinence) throughout the study.
7. Subject is able and willing to comply with study procedures and applicable dressing changes.
8. Subject demonstrates cognitive and physical ability to administer the treatment as determined by the clinician. If a caregiver will administer the treatment, the caregiver must demonstrate cognitive / physical ability.
9. A signed and dated informed consent form has been obtained from the subject.

Exclusion Criteria:

Subjects meeting ANY of the following criteria at time of Screening will be excluded from enrollment:

1. Ulcers with exposed bone or associated with osteomyelitis. Note: Osteomyelitis should be ruled out by clinical examination (probing of the wound) or X-ray findings, if necessary, by the Investigator.
2. Subject has ulcers secondary to a disease other than diabetes, e.g., fungal ulcerations, malignant ulcerations, and ulcerations due to venous or arterial insufficiency, or due to hematological disorders, in the opinion of the Principal Investigator.
3. Ulcer, which in the opinion of the Investigator is suspicious for cancer. Note: Ulcers present for > 6 months would require biopsy to be performed to rule out malignancy.
4. Subjects with a gangrenous or ischemic toe that may need to be amputated in the opinion of the Investigator.
5. Body mass index (BMI) > 40kg/m2
6. Laboratory values at Screening of:

   1. Hemoglobin < 8.5 g/dL
   2. White Blood Cells (WBC) < 3.0 X 109 cells/L and > 11 x 109 cells/L
   3. Liver function studies [Total bilirubin, aspartate aminotransferase (AST) and alanine transaminase (ALT)] > 3x the upper limit of normal
   4. Albumin < 2.5 g/dL
   5. Renal function studies [Serum Creatinine and Urea] > 3x the upper limit of normal
7. Presence of any clinically significant medical condition(s) that, in the opinion of the Investigator, could interfere with wound healing, including but not limited to the following:

   1. Vasculitis or connective tissue disease
   2. Buerger's disease, Raynaud's or other peripheral vascular disease.
   3. Clinically significant claudication or peripheral edema on the affected limb
   4. Acute or unstable Charcot foot
   5. Aplastic anemia or sickle cell anemia
   6. Current sepsis
   7. Severe heart diseases such as congestive heart failure (NYHA Class III or IV), coronary heart disease with ST segment elevation, myocardial infarction, or coronary artery bypass graft or percutaneous transluminal coronary angioplasty within the last 6 months
   8. Severe Liver disease
   9. End-stage renal disease
   10. Severe malnutrition
   11. Immunosuppression
   12. Acquired immune deficiency syndrome (AIDS) or HIV positive
   13. Past or present malignancy below the knee on the same limb as the Target Ulcer;
   14. History of radiation at the Target Ulcer site.
8. Subject is currently receiving (i.e., within 30 days of T1 visit) or scheduled to receive any of following medication or therapies during the course of the study.

   1. immunosuppressants (including chronic systemic corticosteroids)
   2. cytotoxic chemotherapy
   3. cytostatic therapy
   4. Lower limb revascularization surgery (e.g., angioplasty, artery bypass surgery,)
   5. application of bioengineered tissue or skin substitutes
   6. use of any investigational drug(s)
9. Subjects who have previously received NOX1416 treatment
10. Has a known hypersensitivity to any of the investigational drug components
11. Subject is susceptible to hemorrhaging or has a congenital or acquired predisposition to hemorrhaging.
12. Any reason that the subjects may need to be admitted to inpatient acute care in the opinion of the Investigator.
13. Has any other factor which may, in the opinion of the investigator, compromise participation and/or follow-up in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-11-24 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with complete wound closure during the 12 weeks of the Treatment Phase | 12 weeks
  Complete wound closure is defined as 100% re-epithelialization without drainage or dressing requirements confirmed at two consecutive study visits 2 weeks apart. Complete wound closure will be evaluated by the blinded evaluator.

SECONDARY OUTCOMES:
Wound Area Change (%) during the 12 weeks of the Treatment Phase | 12 weeks
  Wound area change is defined as the percentage of wound area change as measured by Swift Imaging device.
Time to complete wound closure during the 12 weeks of the Treatment Phase | 12 weeks
  Complete wound closure was defined as 100% re-epithelialization without drainage or dressing requirements confirmed at two consecutive study visits 2 weeks apart. Complete wound closure will be evaluated by the blinded evaluator.
Frequency of required debridement during the 12 weeks of the Treatment Phase | 12 weeks
  Debridement refers to the process of removing dead/ infected tissue to promote wound healing.
Incidence and severity of treatment-emergent adverse events (TEAEs), including serious adverse events and adverse events resulting in permanent discontinuation of protocol-defined therapy | Up to 24 weeks
  A treatment-emergent adverse event (TEAE) refers to any adverse event that occurs after the first administration of investigational product, i.e., NOX-1416 or the placebo, in this study.
Change in hemoglobin from baseline to subsequent scheduled visits | Up to 24 weeks
  Analysis will be done for Hemoglobin counts.
Change in Hematocrit (HCT) from baseline to subsequent scheduled visits. | Up to 24 weeks
  Analysis will be done for Hematocrit (HCT).
Change in Red Blood Cells (RBC) from baseline to subsequent scheduled visits | Up to 24 weeks
  Analysis will be done for Red Blood Cells (RBC).
Change in White Blood Cells (WBC) from baseline to subsequent scheduled visits | Up to 24 weeks
  Analysis will be done for White Blood Cells (WBC) with total and differential count.
Change in Absolute Neutrophil Counts (ANC) from baseline to subsequent scheduled visits | Up to 24 weeks
  Analysis will be done for levels of Absolute Neutrophil Count (ANC).
Changes in alkaline phosphatase levels in blood from baseline to subsequent scheduled visits | Up to 24 weeks
  Analysis will be done for alkaline phosphatase levels as an indicator of Hepatic function.
Changes in alanine aminotransferase (ALT) levels in blood from baseline to subsequent scheduled visits | Up to 24 weeks
  Analysis will be done for alanine aminotransferase (ALT) as an indicator of Hepatic function.
Changes in total bilirubin levels in blood from baseline to subsequent scheduled visits | Up to 24 weeks
  Analysis will be done for total bilirubin as an indicator of Hepatic function.
Changes in aspartate aminotransferase (AST) levels in blood from baseline to subsequent scheduled visits | Up to 24 weeks
  Analysis will be done for aspartate aminotransferase (AST) as an indicator of Hepatic function.
Changes in total protein levels in blood from baseline to subsequent scheduled visits | Up to 24 weeks
  Analysis will be done for total protein as an indicator of Hepatic function.
Changes in albumin levels in blood from baseline to subsequent scheduled visits | Up to 24 weeks
  Analysis will be done for albumin as an indicator of Hepatic function.
Changes in blood glucose (random) levels from baseline to subsequent scheduled visits | Up to 24 weeks
  Analysis will be done for glucose (random) levels.
Changes in cholesterol (total) levels from baseline to subsequent scheduled visits | Up to 24 weeks
  Analysis will be done for cholesterol (total) levels.
Changes in Lactate dehydrogenase (LDH) levels in blood from baseline to subsequent scheduled visits | Up to 24 weeks
  Analysis will be done for Lactate dehydrogenase (LDH) as an indicator of Hepatic function.
Change in platelets from baseline to subsequent scheduled visits | Up to 24 weeks
  Analysis will be done for platelets levels.
Changes in serum creatinine levels levels in blood from baseline to subsequent scheduled visits | Up to 24 weeks
  Analysis will be done for serum creatinine as an indicator of Renal function.
Changes in urea levels levels in blood from baseline to subsequent scheduled visits | Up to 24 weeks
  Analysis will be done for urea as an indicator of Renal function.
Changes in sodium levels in blood from baseline to subsequent scheduled visits | Up to 24 weeks
  Analysis will be done for electrolytes like sodium.
Changes in potassium levels in blood from baseline to subsequent scheduled visits | Up to 24 weeks
  Analysis will be done for electrolytes like potassium.
Changes in chloride levels in blood from baseline to subsequent scheduled visits | Up to 24 weeks
  Analysis will be done for electrolytes like chloride.
Changes in calcium levels in blood from baseline to subsequent scheduled visits. | Up to 24 weeks
  Analysis will be done for electrolytes like calcium.
Changes in bicarbonate levels in blood from baseline to subsequent scheduled visits | Up to 24 weeks
  Analysis will be done for electrolytes like bicarbonate.
Change in color of urine from baseline to subsequent scheduled visits | Up to 24 weeks
  Urine samples will be tested for their color.
Change in appearance of urine from baseline to subsequent scheduled visits | Up to 24 weeks
  Urine samples will be tested for their appearance.
Change in specific gravity of urine from baseline to subsequent scheduled visits | Up to 24 weeks
  Urine samples will be tested for its specific gravity.
Change in pH of urine specimens from baseline to subsequent scheduled visits | Up to 24 weeks
  Urine samples will be tested for pH levels.
Change in microscopic examination of urine specimens from baseline to subsequent scheduled visits | Up to 24 weeks
  Urine samples will be tested for microscopic examination of urine sediment.
Changes in glucose levels in urine from baseline to subsequent scheduled visits | Up to 24 weeks
  Urine samples will be tested for presence or absence of occult blood.
Change in occult blood in urine samples from baseline to subsequent scheduled visits | Up to 24 weeks
  Urine samples will be tested occult blood.
Changes in ketone levels in urine from baseline to subsequent scheduled visits | Up to 24 weeks
  Urine samples will be tested for ketones.
Changes in leucocyte esterase levels in urine from baseline to subsequent scheduled visits | Up to 24 weeks
  Urine samples will be tested for leucocyte esterase levels.
Changes in nitrite levels in urine from baseline to subsequent scheduled visits | Up to 24 weeks
  Urine samples will be tested for nitrite levels.
Changes in bilirubin levels in urine from baseline to subsequent scheduled visits | Up to 24 weeks
  Urine samples will be tested for bilirubin.
Changes in urobilinogen levels in urine from baseline to subsequent scheduled visits | Up to 24 weeks
  Urine samples will be tested for urobilinogen levels.
Changes in physical examination for general appearance, head, ears, eyes, nose, throat (HEENT) from baseline to subsequent scheduled visits | Up to 24 weeks
  The physical examination will include routine examinations for the following: constitutional/general appearance, head, ears, eyes, nose, throat (HEENT).
Changes in physical examination for cardiovascular parameters from baseline to subsequent scheduled visits | Up to 24 weeks
  The investigator will classify cardiovascular parameters as normal or abnormal. If abnormal, the investigator will specify if the abnormalities are clinically significant or not clinically significant.
Changes in physical examinations for musculoskeletal and extremities from baseline to subsequent scheduled visits | Up to 24 weeks
  The investigator will classify musculoskeletal and extremities parameters as normal or abnormal. If abnormal, the investigator will specify if the abnormalities are clinically significant or not clinically significant.
Changes in physical examinations for dermatologic parameters from baseline to subsequent scheduled visits | Up to 24 weeks
  The investigator will classify dermatologic parameters as normal or abnormal. If abnormal, the investigator will specify if the abnormalities are clinically significant or not clinically significant.
Changes in physical examinations for neurologic parameters from baseline to subsequent scheduled visits | Up to 24 weeks
  The investigator will classify neurologic parameters as normal or abnormal. If abnormal, the investigator will specify if the abnormalities are clinically significant or not clinically significant.
Changes in physical examinations for respiratory parameters from baseline to subsequent scheduled visits | Up to 24 weeks
  The investigator will classify respiratory parameters as normal or abnormal. If abnormal, the investigator will specify if the abnormalities are clinically significant or not clinically significant.
Changes in physical examinations for gastrointestinal parameters from baseline to subsequent scheduled visits | Up to 24 weeks
  The investigator will classify gastrointestinal parameters as normal or abnormal. If abnormal, the investigator will specify if the abnormalities are clinically significant or not clinically significant.
Changes in physical examinations for genitourinary parameters from baseline to subsequent scheduled visits | Up to 24 weeks
  The investigator will classify genitourinary parameters as normal or abnormal. If abnormal, the investigator will specify if the abnormalities are clinically significant or not clinically significant.
Changes in physical examinations for lymphatic parameters from baseline to subsequent scheduled visits | Up to 24 weeks
  The investigator will classify lymphatic parameters as normal or abnormal. If abnormal, the investigator will specify if the abnormalities are clinically significant or not clinically significant.
Changes in physical examinations for psychiatric parameters from baseline to subsequent scheduled visits | Up to 24 weeks
  The investigator will classify psychiatric parameters as normal or abnormal. If abnormal, the investigator will specify if the abnormalities are clinically significant or not clinically significant.
Changes in blood pressure from baseline to subsequent scheduled visits | Up to 24 weeks
  Systolic and diastolic blood pressure will be measured in supine position after subject has been resting for 5 minutes.
Changes in heart rate from baseline to subsequent scheduled visits | Up to 24 weeks
  Heart rate will be measured after subject has been resting for 5 minutes.
Changes in respiratory rate from baseline to subsequent scheduled visits | Up to 24 weeks
  Respiratory rate will be measured in breaths per minute.
Changes in oral temperature from baseline to subsequent scheduled visits | Up to 24 weeks
  Oral temperature will be measured in Fahrenheit.
Changes in Wound-Q Health-Related Quality of Life outcome during the 12 weeks of the Treatment Phase as measured by changes in the subject response to the Wound-Q Health-Related Quality of Life scale | 12 weeks
  The Wound-QoL (Questionnaire on quality of life with chronic wounds) Wound-Q Health-Related Quality of Life assessment includes Life Impact, Psychological and Social scales. The minimum/maximum scores lie between 23 - 92. A lower score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Halperin, MD, Study Chair — Mission Community Hospital, CA
Locations (6):
- Israel (6):
  - Soroka Medical Center (Site 106), Beersheba
  - Carmel Medical Center (Site 104), Haifa
  - Shaare Zedek Hospital (site 101), Jerusalem
  - Hadassah Medical Organization (Site 105), Jerusalem
  - Meir Medical Center (Site 103), Jerusalem
  - Laniado Hospital (Site 102), Netanya

IPD SHARING:
Plan to Share IPD: No